CLINICAL TRIAL: NCT03070249
Title: Compassion Fatigue Among Emergency Department Healthcare Providers
Brief Title: Compassion Fatigue in ED Providers
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201602339
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Compassion Fatigue
Keywords: Emergency Department
MeSH Terms: conditions — Compassion Fatigue; Emergencies | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Emergency Department Healthcare Providers: This study will assess compassion fatigue among healthcare providers in a single emergency department (ED) using the Professional Quality of Life (ProQoL) scale.
  Interventions: Behavioral: Professional Quality of Life (ProQoL) scale

INTERVENTIONS:
Behavioral: Professional Quality of Life (ProQoL) scale — COMPASSION SATISFACTION AND COMPASSION FATIGUE (PROQOL) measures how compassion for those who are cared for can affect providers in positive and negative ways. Questions about experiences, both positive and negative, as a provider reflecting the frequency experiences within the last 30 days. 1=Never 2=Rarely 3=Sometimes 4=Often 5=Very Often

SUMMARY:
This study will assess compassion fatigue among healthcare providers in a single emergency department (ED) using the Professional Quality of Life (ProQoL) scale.

ELIGIBILITY:
Inclusion Criteria:

* Currently employed as a health care provider in the emergency department. All eligible individuals will be 18 years and older.

Exclusion Criteria:

* Individuals that are not currently employed in the emergency department

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is health care providers working in the emergency department.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2017-04-25 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
Assess Compassion Fatigue as precursory research | Baseline
  Professional Quality of Life Scale survey (PROQOL) assesses compassion satisfaction and compassion fatigue. 1=Never 2=Rarely 3=Sometimes 4=Often 5=Very Often

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Carmelle Elie, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No